CLINICAL TRIAL: NCT00288457
Title: Ureteral Stent Length and Patient Symptoms
Status: Terminated | Type: Observational
Why Stopped: Because no staff to consent or enroll subjects
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John G Pattaras, MD, Associate Professor, Emory University
Other Study IDs: 0758-2003
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Ureteral Stent — Ureteral stents are not investigatory but rather part of standard of care. In this study, we were interested in having patients fill out pre and post-operative questionnaires so that we could compare their symptoms with the length of their ureter and the stent placed.

SUMMARY:
The Study of whether or not Ureteral Stent Length affects patient comfort after electro-shock wave treatment for kidney stones.

DETAILED DESCRIPTION:
Patients undergoing electro shock wave for treatment of kidney stones are randomized to long or short stent length after signing an informed consent prior to their surgery. They keep a pain diary and medication diary for a two week period after the stent is placed. These are turned in at the two week post-op visit. Patients also complete a quality of life and urinary symptom score questionnaire pre and post operatively.

ELIGIBILITY:
Inclusion Criteria: Male or female over 18 years of age, will be receiving electro-shock wave therapy for kidney stones -

Exclusion Criteria:Under 18 years of age, inability to give informed consent

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female over 18 years of age, will be receiving electro-shock wave therapy for kidney stones
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2006-02; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John G Pattaras, MD, Principal Investigator — Emory University